CLINICAL TRIAL: NCT04666454
Title: BROKEN-SWEDEHEART- Optimized Pharmacological Treatment for Broken Heart (Takotsubo) Syndrome. A Multinational, Multicentre, Registry-based, Open-label, Randomized Controlled Trial.
Brief Title: BROKEN-SWEDEHEART- Optimized Pharmacological Treatment for Broken Heart (Takotsubo) Syndrome.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BROKEN SWEDEHEART
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Adenosine; Dipyridamole; apixaban; Tablets

STUDY DESIGN:
Intervention Model Description: Multinational, Multicentre, registry-based, open-label, randomized controlled trial with 2 × 2 factorial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Randomisation 1: Adenosine and Dipyridamole (Active Comparator): Adenosine infusion 70 µg/kg/min for 3 hours, followed (first dose 60 minutes apart from the end of the adenosine infusion) by daily oral treatment with the adenosine reuptake inhibitor dipyridamole (200 mg b.i.d.) until normalization of Left Ventricular (LV) function (EF≥50%) is documented on the study-specific echocardiographic assessment at 48-96 hours or at any subsequent echocardiographic examination, or for 30+7 Days.
  Interventions: Drug: Adenosine; Drug: Dipyridamole 200 mg
- Randomisation 1: Control (Other): Care as recommended by the Taskforce on Takotsubo Syndrome of the Heart Failure Association of the European Society of Cardiology.
  Interventions: Other: Care as recommended by the Taskforce on Takotsubo Syndrome of the Heart Failure Association of the European Society of Cardiology for takotsubo syndrome
- Randomisation 2: Apixaban (Active Comparator): Apixaban 5mg b.i.d. per oral until normalization of LV function (EF≥50%) is documented on the study-specific echocardiographic assessment at 48-96 hours or any subsequent echocardiographic examination, or for 30+7 Days.
  Interventions: Drug: Apixaban 5 mg Oral Tablet
- Randomisation 2: No anticoagulant therapy (No Intervention)

INTERVENTIONS:
Drug: Adenosine — Adenosine infusion 70 µg/kg/min for 3 hours.
  Arms: Randomisation 1: Adenosine and Dipyridamole
Drug: Dipyridamole 200 mg — 200 mg b.i.d
  Arms: Randomisation 1: Adenosine and Dipyridamole
Drug: Apixaban 5 mg Oral Tablet — 5mg b.i.d
  Arms: Randomisation 2: Apixaban
Other: Care as recommended by the Taskforce on Takotsubo Syndrome of the Heart Failure Association of the European Society of Cardiology for takotsubo syndrome — This treatment will vary depending on local routines and the degree of adherence to the recommendations.
  Arms: Randomisation 1: Control

SUMMARY:
The aim of this study is to document an optimized pharmacologic treatment for patients with Takotsubo Syndrome. There is currently no published documentation in a large number of patients. The study is a Randomized Registry Clinical Trial and in total 1000 patients registered in SWEDEHEART will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. A clinical diagnosis of TS (see definition 2.1), including an ejection fraction (EF) ˂ 50 % at baseline
3. Written informed consent obtained

Exclusion Criteria:

1. Previous randomization in the trial
2. Any concomitant condition resulting in a life expectancy of less than one month
3. Previously diagnosed left ventricular ejection fraction <50%
4. Known cardiomyopathy (except previous Takotsubo syndrome)
5. Known hemodynamically significant valve disease (moderate or severe aortic/mitral regurgitation) or stenosis
6. Heart transplant or left ventricular assist device recipient
7. Most recent (within the most recent 3 months) haemoglobin ˂10 g/dL
8. Systolic blood pressure <80 mm Hg at screening
9. Estimated glomerular filtration rate <30 mL/min/1.73m2
10. Current dialysis
11. Pregnancy or of childbearing potential who is not sterilized or is not using a medically accepted form of contraception
12. Not suitable in the opinion of the investigator due to severe or terminal comorbidity with poor prognosis, or characteristics that may interfere with adherence to the trial protocol

    Specific exclusion criteria for Randomization 1
13. Any contra-indication for treatment with adenosine or dipyridamole (including AV-block II and III, sick-sinus syndrome in subjects who don´t have a functioning pacemaker, unstable angina, ongoing treatment with dipyridamole)
14. Severe asthma (defined as asthma requiring medium or high-dose inhaled corticosteroids combined with other long-acting medications) and severe Chronic Obstructive Pulmonary Disease (COPD), (defined as FEV-1 ˂ 50 %)
15. Ongoing treatment with dipyridamole
16. Declined participation in study 1

Specific exclusion criteria for Randomization 2

1. Any contra-indication for anticoagulant treatment.
2. Current indication for treatment with, anticoagulant or dual antiplatelet therapy
3. Declined participation in study 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Randomization 1: First co-primary endpoint: Wall motion score index (defined as the semi-quantitative score according to the American Society of Echocardiography) | 48-96 hours
Randomization 1: Second co-primary endpoint: The occurrence of the composite of death, cardiac arrest, or the need for cardiac mechanical assist device, or re-hospitalization for heart failure or ejection fraction <50% | up until day 30 day respectively at 48-96 hours
Randomization 2: The occurrence of any thromboembolic event (defined as ischemic stroke, peripheral arterial embolization or myocardial infarction) or death, or the presence of a cardiac thrombus, as assessed by echocardiography | up until day 30 respectively 48-96 hours

SECONDARY OUTCOMES:
Randomization 1: The hierarchical occurrence (in descending order of importance) of time to death, time to cardiac assist device, time to cardiac arrest and ejection fraction <50% | all time to the first occurrence up until day 30 respectively at 48-96 hours (binary)
Randomization 1: Ejection fraction | at 48-96 hours (continuous)
Randomization 1: Any sustained ventricular tachycardia or fibrillation | within 48-96 hours (binary)
Randomization 1: Any high-grade atrioventricular block or sinus arrest | within 48-96 hours (binary)
Randomization 1: Need for cardiac assist device | up until day 30 day (binary)
Randomization 1: Death | up until day 30 (binary)
Randomization 1: Stroke | up until day 30 (binary)
Randomization 1: Worsening heart failure in hospital (defined as worsening signs or symptoms of heart failure, necessitating intensification of intravenous pharmacologic heart failure therapy or mechanical ventilation) | up until day 30
Randomization 2: Presence of cardiac thrombus | at 48-96 hours
Randomization 2: Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria minor or major | up until day 30 (binary)
Randomization 2: Bleeding Academic Research Consortium (BARC) grade 2-5 | up until day 30 (binary)
Randomization 2: BARC grade 3-5 | up until day 30 (binary)
Randomization 2: Any blood transfusion | up until day 30 (binary)

CONTACTS AND LOCATIONS:
Overall Officials: Elmir Omerovic, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (16):
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
- Oslo University Hospital, Oslo, Norway
- Sweden (13):
  - Östersund Sjukhus, Östersund, Jämtland Härjedalen
  - Region Jönköpings Län, Jönköping, Region Jönköping
  - Norra Älvsborgs länssjukhus, Trollhättan, Västra Götalands Region
  - Region Dalarna, Falun
  - Sahlgrenska University Hospital, Department of Cardiology, Gothenburg
  - Skaraborg Hospital, Gothenburg
  - Region Skane Helsingborg Hospital, Helsingborg
  - Region Oestergoetland, Linköping
  - Region Skane - Skanes Universitetssjukhus, Lund
  - Region Orebro lan, Örebro
  - Danderyds Hospital, Department of Cardiology, Stockholm
  - Karolinska University Hospital, Huddinge, Department of Cardiology, Stockholm
  - Umeå University Hospital, Department of Cardiology, Umeå

IPD SHARING:
Plan to Share IPD: Yes
To be decided.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: To be decided
Access Criteria: To be decided (TBD)

REFERENCES:
- [Derived] Omerovic E, James S, Erlinge D, Hagstrom H, Venetsanos D, Henareh L, Ekenback C, Alfredsson J, Hambreus K, Redfors B. Rationale and design of BROKEN-SWEDEHEART: a registry-based, randomized, parallel, open-label multicenter trial to test pharmacological treatments for broken heart (takotsubo) syndrome. Am Heart J. 2023 Mar;257:33-40. doi: 10.1016/j.ahj.2022.11.010. Epub 2022 Nov 23. PMID 36435233